CLINICAL TRIAL: NCT06987695
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Maridebart Cafraglutide in Adult Participants in Japan Who Have Obesity Disease (MARITIME 3-J)
Brief Title: Efficacy and Safety of Maridebart Cafraglutide in Adult Participants in Japan Who Have Obesity Disease
Acronym: MARITIME-3-J
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20230144
Record Dates: First submitted 2025-05-02; First posted 2025-05-23 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Obesity Disease
Keywords: Overweight; BMI; Body weight; Maridebart cafraglutide; Chronic weight management; MariTide; Type 2 Diabetes Mellitus; T2DM
MeSH Terms: conditions — Overweight; Body Weight; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Maridebart Cafraglutide High Dose (Experimental): Participants will receive maridebart cafraglutide high dose subcutaneously (SC) for 72 weeks.
  Interventions: Drug: Maridebart cafraglutide
- Maridebart Cafraglutide Medium Dose (Experimental): Participants will receive maridebart cafraglutide medium dose SC for 72 weeks.
  Interventions: Drug: Maridebart cafraglutide
- Maridebart Cafraglutide Low Dose (Experimental): Participants will receive maridebart cafraglutide low dose SC for 72 weeks.
  Interventions: Drug: Maridebart cafraglutide
- Placebo (Placebo Comparator): Participants will receive placebo SC for 72 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Maridebart cafraglutide — Maridebart cafraglutide will be administered SC.
  Other Names: AMG 133; MariTide
  Arms: Maridebart Cafraglutide High Dose; Maridebart Cafraglutide Low Dose; Maridebart Cafraglutide Medium Dose
Drug: Placebo — Placebo will be administered SC.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to demonstrate that maridebart cafraglutide is superior to placebo for percent change in body weight and proportion of participants with ≥ 5% reduction in body weight.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* History of at least 1 self-reported unsuccessful attempt at weight loss by diet and exercise.
* Body mass index (BMI) ≥ 35 kg/m^2 at screening with a current diagnosis of at least 1 of the weigh-related comorbidities specified in the Japan Society for the Study of Obesity (JASSO) guideline OR BMI ≥ 27 kg/m^2 to < 35 kg/m^2 at screening, with a current diagnosis of at least 2 of the weight-related comorbidities specified in the JASSO guideline.
* For both BMI categories, at least 1 of the weight-related comorbidities must be hypertension, dyslipidemia, or T2DM according to the definitions below:

  1. hypertension: treated, or with SBP ≥ 140 mmHg, or DBP ≥ 90 mmHg at screening.
  2. dyslipidemia: treated, or with LDL > 140 mg/dL (3.6 mmol/L), or triglycerides ≥ 150 mg/dL (1.7 mmol/L), or non-HDL cholesterol > 170 mg/dL (4.4 mmol/L) or HDL < 40 mg/dL (1.0 mmol/L) at screening.
  3. T2DM: diagnosed ≥ 180 days before screening, and treated with diet and exercise alone and/or a stable treatment for at least 90 days before screening with up to 3 oral glucose-lowering medications (as per local labeling) (except for glucagon-like peptide-1 receptor agonists [GLP-1RA] and dipeptidyl peptidase-4 [DPP-4] inhibitors), and have a HbA1c ≥ 7% and ≤ 10% (53-86 mmol/mol) at screening.
* In the opinion of the investigator, well-motivated and willing to:

  1. Follow study procedures for the duration of the study, including, but not limited to, follow lifestyle advice, maintain a study log(s)/diary(ies), and complete required study visits and questionnaires.
  2. Perform self-monitoring blood glucose (SMBG) per protocol (only for participants with T2DM).

Exclusion Criteria:

* Obesity induced by other endocrinological disorders or monogenetic or syndromic forms of obesity.
* Self-reported change in body weight > 5 kg within 90 days before screening.
* Previous or planned (during the study) surgical, endoscopic, or device-based treatment for obesity.
* For participants without diabetes at screening, type 1 or 2 diabetes mellitus or any other types of diabetes mellitus (except history of gestational diabetes).
* For participants with T2DM at screening, any other type(s) of diabetes mellitus except T2DM.
* History of chronic pancreatitis or history of acute pancreatitis within 180 days before screening.
* Family (first-degree relative[s]) or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN-2).
* History of unstable major depressive disorder (MDD) or other severe psychiatric disorder within 2 years before screening.
* Lifetime history of suicide attempt.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2025-06-13 (Actual); Primary Completion 2027-04-27 (Estimated); Study Completion 2027-07-21 (Estimated)

PRIMARY OUTCOMES:
Percent Change From Baseline in Body Weight at Week 72 | Baseline and Week 72
Participants Achieving ≥ 5% Reduction in Body Weight From Baseline at Week 72 | Baseline and Week 72

SECONDARY OUTCOMES:
Change From Baseline in Waist Circumference at Week 72 | Baseline and Week 72
Participants Achieving ≥ 10% Reduction in Body Weight from Baseline at Week 72 | Baseline and Week 72
Participants Achieving ≥ 15% Reduction in Body Weight from Baseline at Week 72 | Baseline and Week 72
Change From Baseline in Body Weight at Week 72 | Baseline and Week 72
Percent Change From Baseline in Body Weight in Participants Without Type 2 Diabetes Mellitus (T2DM) at Week 72 | Baseline and Week 72
Percent Change From Baseline in Body Weight in Participants With T2DM at Week 72 | Baseline and Week 72
Change From Baseline in Body Mass Index (BMI) at Week 72 | Baseline and Week 72
Participants Achieving ≥ 20% Reduction in Body Weight from Baseline at Week 72 | Baseline and Week 72
Change From Baseline in Visceral Fat Area (VFA) at Week 72 | Baseline and Week 72
Participants Achieving VFA < 100 cm^2 in VFA at Week 72 | Week 72
Percent Change From Baseline in Fasting Total Cholesterol at Week 72 | Baseline and Week 72
Percent Change From Baseline in Fasting Non-high-density Lipoprotein Cholesterol (non-HDL-C) at Week 72 | Baseline and Week 72
Percent Change From Baseline in Fasting Low-density Lipoprotein Cholesterol (LDL-C) at Week 72 | Baseline and Week 72
Percent Change From Baseline in Fasting Triglycerides at Week 72 | Baseline and Week 72
Percent Change From Baseline in Fasting Very Low-density Lipoprotein Cholesterol (VLDL-C) at Week 72 | Baseline and Week 72
Percent Change From Baseline in Fasting High-density Lipoprotein Cholesterol (HDL-C) at Week 72 | Baseline and Week 72
Change From Baseline in Systolic Blood Pressure (SBP) at Week 72 | Baseline and Week 72
Change From Baseline in Diastolic Blood Pressure (DBP) at Week 72 | Baseline and Week 72
Change From Baseline in Fasting Plasma Glucose at Week 72 | Baseline and Week 72
Percent Change From Baseline in Fasting Insulin at Week 72 | Baseline and Week 72
Change from Baseline in Hemoglobin A1c (HbA1c) at Week 72 | Baseline and Week 72
Percentage of Participants with a Change from Baseline in Glycemic Status at Week 72 for Participants Without T2DM at Baseline | Baseline and Week 72
  Glycemic status was categorized as:
  * normoglycemic (fasting plasma glucose < 100 mg/dL and HbA1c < 5.7%, in absence of T2DM diagnosis),
  * prediabetes (fasting plasma glucose 100 - 125 mg/dL or HbA1c 5.7% - 6.4% in the absence of a T2DM diagnosis),
  * or, T2DM (fasting plasma glucose ≥ 126 mg/dL and HbA1c ≥6.5%).
Participants With T2DM Achieving HbA1c < 7% at Week 72 | Week 72
Participants With T2DM Achieving HbA1c ≤ 6.5% at Week 72 | Week 72
Participants With T2DM Achieving HbA1c < 5.7% at Week 72 | Week 72
Change From Baseline in Short Form 36 Health Survey Version 2 (SF-36v2) Acute Physical Function Domain Score at Week 72 | Baseline and Week 72
  The SF-36v2 Acute Physical Function domain score measures an individual's ability to perform daily physical activities, such as walking and climbing stairs, over the past week. It includes 10 items scored on a 3-point Likert scale, with raw scores transformed to a 0-100 scale. Higher scores indicate better physical functioning and fewer limitations due to physical health.
Change from Baseline in the Impact of Weight on Quality of Life-Lite Clinical Trials Version (IWQOL-Lite-CT) Physical Function Composite Score at Week 72 | Baseline and Week 72
  The IWQOL-Lite-CT is a 20-item questionnaire designed to assess the impact of weight on quality of life in clinical trials. Items are scored on a 5-point Likert scale, with raw scores transformed to a 0-100 scale, where higher scores indicate better quality of life and less weight-related impact.
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Up to Week 84
Number of Participants Experiencing Serious Adverse Events | Up to Week 84
Plasma Concentration of Maridebart Cafraglutide at Week 72 | Week 72

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (30):
- Japan (30):
  - Meitetsu Hospital, Nagoya, Aichi-ken
  - Hosokawa Surgical Clinic, Nagoya, Aichi-ken
  - Social Medical Corporation Kojunkai Daido Clinic, Nagoya, Aichi-ken
  - Wellness Tenjin Clinic, Fukuoka, Fukuoka
  - Medical Corporation Boocs Boocs Clinic Fukuoka, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Tashiro Endocrinology Clinic, Fukuoka, Fukuoka
  - Fukuoka Shinmizumaki Hospital, Onga-gun, Fukuoka
  - Matsunami Health Promotion Clinic, Hashima-gun, Gifu
  - Manda Memorial Hospital, Sapporo, Hokkaido
  - Yamasaki Family Clinic, Amagasaki-shi, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - Deguchi Clinic, Kobe, Hyōgo
  - Nishiyamado Keiwa Hospital, Naka, Ibaraki
  - Aira Diabetes Thyroid Internal Medicine Clinic, Aira-shi, Kagoshima-ken
  - Matsuba Clinic, Kawasaki-shi, Kanagawa
  - Medical Corporation Keiseikai Kajiyama Clinic, Kyoto, Kyoto
  - Kyoto University Hospital, Kyoto, Kyoto
  - Midori Clinic, Nagasaki, Nagasaki
  - Urasoe General Hospital, Urasoe-shi, Okinawa
  - Joh Medical Clinic, Osaka, Osaka
  - Adachi Kyosai Hospital, Adachi-ku, Tokyo
  - Nihonbashi Sakura Clinic, Chuo-ku, Tokyo
  - Medical Corporation Chiseikai Tokyo Center Clinic, Chuo-ku, Tokyo
  - Medical Corporation Kenshinkai Minamino Cardiovascular Hospital, Hachioji-shi, Tokyo
  - Tokyo Saiseikai Central Hospital, Minato-ku, Tokyo
  - Shimamura Memorial Hospital, Nerima-ku, Tokyo
  - MIH Clinic Yoyogi, Shibuya-ku, Tokyo
  - Shinjuku Southern Clinic, Shinjuku-ku, Tokyo
  - Ikebukuro Metropolitan Clinic, Toshima-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com